CLINICAL TRIAL: NCT04280757
Title: Ambispective Comparative Cohort Study to Assess the Differences in Development and Growth Patterns of Biopsied and Non-Biopsied ICSI Embryos and Natural Pregnancy Embryos[BNB-ICSI Study]
Brief Title: Comparison Between Biopsied and Non-biopsied Intracytoplasmatic Sperm Injection (ICSI) Embryos and Natural Pregnancy Embryos
Acronym: BNB-ICSI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wael Elbanna Clinic (Other)
Collaborators: Fetal Medicine Research Center, Spain (Other)
Responsible Party: Principal Investigator, Wael Elbanna, European board fellow of obstetrics and gynecology, Wael Elbanna Clinic
Other Study IDs: Elbanna_2020_02
Record Dates: First submitted 2020-02-10; First posted 2020-02-21 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Women Conceiving by: 1- ICSI-PGS 2- ICSI-non-PGS 3- Spontaneously Conceiving Women
Keywords: fetal growth; biochemical parameters
MeSH Terms: interventions — Phosphatidylglycerols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Arm 1: Biopsied ICSI embryos
  Interventions: Procedure: Biopsied ICSI embryos (PGS)
- Arm 2: Non biopsied ICSI embryos
- Arm 3: Natural pregnancy embryos

INTERVENTIONS:
Procedure: Biopsied ICSI embryos (PGS) — Biopsied ICSI embryos (PGS)
  Groups: Arm 1

SUMMARY:
As Pre Implantation Genetic Screening (PGS) becomes now a replacement modality and trend gaining popularity among physicians and patients on claiming its ability to settle on the simplest genetically normal embryo, so it had been logical to review if taking cells from the embryo in its early development will or won't affect its growth as compared to the previous standard technique of ICSI and in comparison to a normally conceived embryos the study also will question if the parameters of the prenatal biochemical standard parameters will have any differences if the embryo is already genetically tested embryo and compare these parameters with non PGS embryos and normally conceived embryos.

This study is an ambispective, comparative, cohort, observational, single-center study.

The study participants' relevant medical records will be collected and reviewed for the retrospective subjects and after obtaining informed consent for the prospective subjects. The study materials that will be used will include blood tests and ultrasound. The study will involve three study arms

DETAILED DESCRIPTION:
This study is an ambispective, comparative, cohort, observational, single-center study that will be conducted at Wael ElBanna Clinic, a private center that is well equipped for all procedures needed for ICSI and fetal medicine. After obtaining informed consent, the study participants' relevant medical records will be collected and reviewed. Data will be collected from the subjects' medical records. Data will be pooled and presented in aggregate, without identification of individual subjects.

The study materials that will be used will include blood tests and ultrasound. The study will involve three study arms:

* Arm 1: biopsied ICSI embryos (PGS)
* Arm 2: none biopsied ICSI embryos
* Arm 3: natural pregnancy embryos

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnant women
2. Pregnancy confirmation by ultrasound at week 6 of gestation either by normal pregnancy or ICSI (Biopsied and Non-Biopsied)
3. Between the age of 20 and 40 years.
4. Non-smokers.
5. BMI must be between 19 and 40

Exclusion Criteria:

1. Those with anti-phospholipid syndrome confirmed by serological tests
2. Those with any hematological and immunological disorders
3. Women with uterine abnormalities have not been corrected.
4. Women with systemic diseases that cannot be controlled or managed

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: The study population include women conceiving by:
  1. ICSI-PGS
  2. ICSI-non-PGS
  3. Spontaneously conceiving women
Sampling Method: Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
First primary endpoint | At pregnancy
  - Early ultrasound measurements "yolk sac (YS), mean sac diameter (MSD), crown rump length (CRL)", different maternal serum prenatal screening markers for growth and aneuploidy between the three arms* of the study
Second primary endpoint | At 2nd trimester of pregnancy
  - Second trimetric U/S measurements of fetal growth : U/S measurements of fetal growth using growth curves and measurement of FPI (fetal ponderal index) and fetal weight percentile
Third primary endpoint | At 3rd trimester of pregnancy
  - Third-trimester U/S measurements of fetal growth : U/S measurements of fetal growth using growth curves and measurement of FPI (fetal ponderal index) and fetal weight percentile

SECONDARY OUTCOMES:
First secondary endpoint | At Labor
  Miscarriage
Second secondary endpoint | At Labor
  Live-birth weight
Third secondary endpoint | At Labor
  Preterm labor

CONTACTS AND LOCATIONS:
Overall Officials: Wael Elbanna, Specialist, Study Director — Wael Elbanna Clinic; Eduard Gratacos, Specialist, Principal Investigator — fetal medicine; Manal El-Hinnawi, Specialist, Principal Investigator — Wael Elbanna Clinic
Locations (1):
- wael Elbanna Clinic, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided